CLINICAL TRIAL: NCT06808139
Title: Pearls and Pitfalls in Usage of Plasma-Rich Platelet Graft Versus Dartos Flap in Distal Penile Hypospadias Repair
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed ali amen diab, residant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRPgraft/DartosflapHypospadias
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Penile Hypospadias
Keywords: Plasma-Rich Platelet Graft; Dartos Flap
MeSH Terms: conditions — Hypospadias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): Plasma-Rich Platelet Graft
  Interventions: Procedure: Plasma-Rich Platelet Graft
- Group B (Active Comparator): Dartos Flap
  Interventions: Procedure: Dartos Flap

INTERVENTIONS:
Procedure: Plasma-Rich Platelet Graft — The clot was extracted from the tube, separated from red blood cells, and gently compressed between two surgical swabs to obtain a soft and resistant membrane. The Snodgrass technique was carried out for all patients, with a suitable size catheter (8-12-Fr), repair was carried out by a continuous layer of polyglycolic suture (Vicryl) size 6/0, covered by an interrupted second layer. In group A, after finishing the Snodgrass TIPU, a PRP sheet coverage was applied over urethroplasty and secured by Vicryl 7/0, and finally the skin sutured directly without any covering layers
  Arms: Group A
Procedure: Dartos Flap — preputial dartos flap will be used
  Arms: Group B

SUMMARY:
Hypospadias is the most common congenital anomaly of penis. It is the second most common genital birth defect in boys after cryptorchidism The reinforcement of hypospadias repair with an intermediate layer is believed to reduce the incidence of postoperative complications such as uretherocautanous fistula.

Hypospadias is classified by the location of the abnormal urethral meatus into distal penile (glandular ,subcoronal and distal penile), mid penile and proximal penile hypospadias Indeed, uretherocautanous fistula is most common complication after urethroplasty, with introduction of a protective layer between the neourethra and the covering skin strongly reduces fistulas occurrence and the overall complication the aim of the study To evaluate and to compare the use of PRP covering layer and dartos fascia flap layer in regard to complication rates in hypospadias repair

DETAILED DESCRIPTION:
Hypospadias is the most common congenital anomaly of penis. It is the second most common genital birth defect in boys after cryptorchidism The reinforcement of hypospadias repair with an intermediate layer is believed to reduce the incidence of postoperative complications such as uretherocautanous fistula.

Hypospadias is classified by the location of the abnormal urethral meatus into distal penile (glandular ,subcoronal and distal penile), mid penile and proximal penile hypospadias Indeed, uretherocautanous fistula is most common complication after urethroplasty, with introduction of a protective layer between the neourethra and the covering skin strongly reduces fistulas occurrence and the overall complication the aim of the study To evaluate and to compare the use of PRP covering layer and dartos fascia flap layer in regard to complication rates in hypospadias repair

ELIGIBILITY:
Inclusion Criteria:

* Age >6 months
* Distal penile hypospadias
* Denovo hypospadias

Exclusion Criteria:

* Recurrent hypospadias -Mid and proximal penile hypospadias

Min Age: 6 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male
Enrollment: 70 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
incidence of occurrence of uretherocutanous fistula | 6 month
  occurrence of conection between urthera and skin

IPD SHARING:
Plan to Share IPD: Undecided